CLINICAL TRIAL: NCT03923049
Title: Feasibility and Accuracy of Hybrid Magnetic Resonance and Positron Emission Tomography With 18F-Fluorodeoxyglucose in Diagnosing Cardiac Sarcoidosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and support
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Navkaranbir Bajaj, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300002877
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MRI (Other): Diagnostic testing with simultaneous PET/MRI for cardiac sarcoidosis diagnosis
  Interventions: Diagnostic Test: hybrid PET/MRI

INTERVENTIONS:
Diagnostic Test: hybrid PET/MRI — On the day of the procedure, subjects will undergo a PET scan followed by MRI scan.

SUMMARY:
The purpose and objectives of the study is to establish the feasibility of the simultaneous PET/MR in patients with cardiac sarcoidosis, determine relationships between various imaging biomarkers like extracellular volume (ECV) and standardized uptake values (SUV) from FDG-PET and to evaluate the diagnostic accuracy of the simultaneous method in comparison to the PET/CT and cardiac MRI.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria and agree to the study will be recruited from the Kirklin Clinic and UAB hospitals who will be undergoing FDG-PET/CT for cardiac study as part of their standard of care to diagnose cardiac sarcoidosis. MRI and FDG-PET screening questionnaire will be completed. A chart review will be completed to obtain data from patient medical records pertaining to study including age, gender, race, weight, height, vital signs, social and family history, past medical history especially if there is any history of hypertension, diabetes, high cholesterol levels, heart failure or history of lung diseases, lab results including brain natriuretic peptide levels, creatinine, hemoglobin, coagulation parameters, results of stress test/left heart catheterization, prior echocardiography if available. The CMR will be done solely for research purposes. The patient will be in the PET/MRI scanner for cardiac study only for 60-90 minutes, Finally, multi-sequence, multi-planar cardiac MR images will be acquired to assess cardiac chamber size, regional wall motion abnormalities, ejection fraction, left ventricular perfusion(using gadolinium-based agent) and late gadolinium enhancement.

The investigators will also conduct MRI examinations on 5 healthy volunteers to establish cardiac MRI protocol for the PET/MRI scanner. These scans will not involve any FDG administration to the healthy volunteers. These will involve cardiac MRI examinations to determine the feasibility and quality of MRI scans with the new scanner.

ELIGIBILITY:
Inclusion Criteria:

1.Subjects older than 18 years of age with high suspicion of cardiac sarcoidosis and/or biopsy proven extracardiac sarcoidosis and/or positive HRS criteria will be enrolled.

Exclusion Criteria:

1. Coronary artery disease
2. Insulin dependent diabetes
3. Claustrophobia
4. Pregnancy/nursing
5. Presence of pacemaker or automatic implantable cardioverter-defibrillator
6. Impaired renal function (estimated glomerular filtration rate <45 ml/min/1.73 m2) will be excluded.
7. Inability to undergo PET/MRI due to any other condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
diagnosing cardiac sarcoidosis using combined 18F-FDG-PET/MRI examination | baseline through 24 hours
  diagnostic accuracy of FDG-PET/MRI test will be determined by comparing the PET/MRI test against the Heart Rhythm Society (HRS) criteria which is the standard of reference.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03923049/ICF_000.pdf